CLINICAL TRIAL: NCT05272111
Title: Effects of Fasciatherapy Versus Facial Manipulation on Pain, Range of Motion and Function in Patients With Chronic Neck Pain
Brief Title: Effects of Fascia Therapy Versus Facial Manipulation on Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCRS/22/0102 Aiman
Record Dates: First submitted 2022-02-20; First posted 2022-03-09 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Neck Pain
Keywords: Neck Pain; Fascia Therapy; Facial Manipulation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia Therapy (Experimental): Group A will receive Fascia therapy
  Interventions: Other: DBM fasciatherapy+ conventional physical therapy
- Facial Manipulation (Experimental): Group B will receive Facial manipulation
  Interventions: Other: fascial manipulation+ conventional physical therapy

INTERVENTIONS:
Other: DBM fasciatherapy+ conventional physical therapy — DBM fasciatherapy (3 sessions per day). It soft, deep and non-manipulative form of treatment that involves the application of gentle pressure while stretching the body's connective tissue. A specialized form of touch, somatic sense, and specific body movement protocols are the three steps involved in the fasciatherapy. + hot pack (10 min) + neck isometrics (neck flexion, extension, side bending) + neck stretches (neck flexors, extensors, side benders and rotation). A total of 45 min session three times a week on alternate days for three weeks
  Arms: Fascia Therapy
Other: fascial manipulation+ conventional physical therapy — Fascial manipulation (3 sessions per day). This technique involves the identification of specific, localized areas of the fascia with limited movements. Once it is identified, then a specific point on the fascia is targeted and through the appropriate manipulation of this precise part of the fascia, movement can be restored. + hot pack (10 min) + neck isometrics (neck flexion, extension, side bending) + neck stretches (neck flexors, extensors, side benders and rotation). A total of 45 min session three times a week on alternate days for three weeks
  Arms: Facial Manipulation

SUMMARY:
This study a randomized clinical trial to determine the effects of fasiatherapy versus facial manipulation on pain, range of motion and function in patients with chronic neck pain. A sample of 52 patients will be taken and divided into two groups each with 26 patients. Group A will receive DBM fasciatherapy along with conventional physical therapy while group B will receive fascial manipulation along with the conventional physical therapy protocol. The conventional physical therapy protocol will include hot pack, neck isometrics and stretches. The session will be around 45 to 60 min on each patient with three session per week on alternate days. A total of three-week treatment regime will be given to the patients and assessment of patient's pain, range of motion and function with NPRS (numeric pain rating scale), goniometry and NDI (neck disability index) will be done at the baseline, after the completion of treatment at three weeks and after 6 weeks to observe the long-term effects. The data will be analyzed using SPSS.

DETAILED DESCRIPTION:
Chronic neck pain is one of the most common musculoskeletal disorder among general population. Like muscular spasm of neck that can cause neck pain, fascial adhesions are also the common cause of neck pain. Fascia is a form of connective tissue that is made up of collagen, surrounds the body parts and also resist tissue tensile load. Fascial injury and adhesions are common and can lead to pain, restricted motion and swelling. The treatment of the fascial injury is necessary to relieve those symptoms. There are many treatments for the chronic neck pain and this study focuses on two new treatment techniques for the fascial pain. The first is the Dannis Bois method fasciatherpy which is a manual approach that focuses on the structural segmentation of fascia and involves the application of gentle pressure while stretching the body's connective tissues. The other treatment technique is the fascial manipulation method that involves the treatment which is directed to specific fascial adhesions. The current study is novel in a way that there is limited literature about DBM fasciatherapy versus fascial manipulation on chronic neck pain. Both methods were employed to see if they improve ranges along with accompanying pain and disability.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Age 18-40 years
* Chronicity of pain - 6 months minimum

Exclusion Criteria:

* Post-op patient
* Any bony, soft tissue or systemic disease
* Pregnant females
* Radiculopathy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2022-02-20 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
1. NPRS (numeric pain rating scale) | 6th Week
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10) that best reflects the intensity of his/her pain 11-point numeric scale ranges from '0' representing no pain to 10 representing the worst imaginable pain.
2. Goniometer | 6th Week
  The science of measuring the joint ranges in each plane of the joint is called goniometry. Goniometer is a device that measures an angle or permits the rotation of an object to a definite position. Neck flexion, extension, side bending and rotation will be assessed through it.
NDI | 6th Week
  The NDI has become a standard instrument for measuring self-rated disability due to neck pain. Each of the 10 items scores from 0 to 5. The maximum score is 50.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, Study Director — Riphah International University; Syeda Aiman Batool, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McLean SM, May S, Klaber-Moffett J, Sharp DM, Gardiner E. Risk factors for the onset of non-specific neck pain: a systematic review. J Epidemiol Community Health. 2010 Jul;64(7):565-72. doi: 10.1136/jech.2009.090720. Epub 2010 May 12. PMID 20466711
- [Background] Quere N, Noel E, Lieutaud A, d'Alessio P. Fasciatherapy combined with pulsology touch induces changes in blood turbulence potentially beneficial for vascular endothelium. J Bodyw Mov Ther. 2009 Jul;13(3):239-45. doi: 10.1016/j.jbmt.2008.06.012. Epub 2008 Aug 12. PMID 19524848
- [Background] Branchini M, Lopopolo F, Andreoli E, Loreti I, Marchand AM, Stecco A. Fascial Manipulation(R) for chronic aspecific low back pain: a single blinded randomized controlled trial. F1000Res. 2015 Nov 3;4:1208. doi: 10.12688/f1000research.6890.2. eCollection 2015. PMID 26834998
- [Background] Rodriguez-Huguet M, Rodriguez-Almagro D, Rodriguez-Huguet P, Martin-Valero R, Lomas-Vega R. Treatment of Neck Pain With Myofascial Therapies: A Single Blind Randomized Controlled Trial. J Manipulative Physiol Ther. 2020 Feb;43(2):160-170. doi: 10.1016/j.jmpt.2019.12.001. Epub 2020 Apr 18. PMID 32317109
- [Background] Mawdsley RH, Moran KA, Conniff LA. Reliability of two commonly used pain scales with elderly patients. Journal of Geriatric Physical Therapy. 2002;25(3):16.
- [Background] Young IA PT, DSc, Dunning J PT, DPT, Butts R PT, PhD, Mourad F PT, DPT, Cleland JA PT, PhD. Reliability, construct validity, and responsiveness of the neck disability index and numeric pain rating scale in patients with mechanical neck pain without upper extremity symptoms. Physiother Theory Pract. 2019 Dec;35(12):1328-1335. doi: 10.1080/09593985.2018.1471763. Epub 2018 Jun 1. PMID 29856244
- [Background] Day JA, Stecco C, Stecco A. Application of Fascial Manipulation technique in chronic shoulder pain--anatomical basis and clinical implications. J Bodyw Mov Ther. 2009 Apr;13(2):128-35. doi: 10.1016/j.jbmt.2008.04.044. Epub 2008 Jun 24. PMID 19329049
- [Background] Courraud C, Bertrand I, Dupuis C. Assessment of the effects of DBM fasciatherapy on fascial system with elastography.
- [Background] Stecco C, Day JA. The fascial manipulation technique and its biomechanical model: a guide to the human fascial system. Int J Ther Massage Bodywork. 2010 Mar 17;3(1):38-40. doi: 10.3822/ijtmb.v3i1.78. No abstract available. PMID 21589701
- [Derived] Batool SA, Shakil-Ul-Rehman S, Tariq Z, Ikram M. Effects of fasciatherapy versus fascial manipulation on pain, range of motion and function in patients with chronic neck pain. BMC Musculoskelet Disord. 2023 Oct 5;24(1):789. doi: 10.1186/s12891-023-06769-0. PMID 37798756